CLINICAL TRIAL: NCT00695318
Title: A Randomized, Double-Masked, Fellow-Eye Comparison Of The Safety And Efficacy Of 0.2 And 0.5 µg/Day Fluocinolone Acetonide Intravitreal Insert To Sham Injection In Subjects With Bilateral Geographic Atrophy Due To AMD
Brief Title: Fluocinolone Acetonide Intravitreal Inserts in Geographic Atrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-01-08-004
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Age-Related Macular Degeneration; Geographic Atrophy; GA
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 2, I 0.2 µg/Day + Sham (Experimental): 0.2 µg/Day
  Interventions: Drug: Fluocinolone Acetonide
- A, 2, II 0.5 µg/Day + Sham (Experimental): 0.5 µg/Day
  Interventions: Drug: Fluocinolone Acetonide

INTERVENTIONS:
Drug: Fluocinolone Acetonide — 0.2 µg/Day in study eye + Sham in fellow eye
  Arms: A, 2, I 0.2 µg/Day + Sham
Drug: Fluocinolone Acetonide — 0.5 µg/Day in study eye +Sham in fellow eye
  Arms: A, 2, II 0.5 µg/Day + Sham

SUMMARY:
This study will compare the safety and efficacy of Medidur FA treatment in one eye to the sham-treated fellow eye of subjects with geographic atrophy secondary to AMD.

DETAILED DESCRIPTION:
Each patient received a sham injection in one eye and active treatment in the other eye. The eye receiving active treatment was selected based on a randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis bilateral GA secondary to AMD of ≥ 0.5 and ≤ 7 MPS disc areas
* Males and non-pregnant females 55 years old or older

Exclusion Criteria:

* GA secondary to any condition other than AMD in either eye
* History of or current CNV in either eye or the need for anti-angiogenic therapy
* Glaucoma or ocular hypertension (IOP > 21 mmHg OR concurrent therapy at screening with IOP-lowering agents) in either eye
* Treatment with intravitreal, subtenon, or periocular steroid within 6 months prior to enrollment in either eye
* Any change in systemic steroid therapy within 3 months of screening
* History of vitrectomy in either eye
* Any ocular surgery within 12 weeks of screening in either eye

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-12; Primary Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kresge Eye Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A, 2, I 0.2 µg/Day + Sham: 0.2 µg/Day
  Fluocinolone Acetonide: 0.2 µg/Day
- A, 2, II 0.5 µg/Day + Sham: 0.5 µg/Day
  Fluocinolone Acetonide: 0.5 µg/Day
Period: Overall Study
Arm/Group | A, 2, I 0.2 µg/Day + Sham | A, 2, II 0.5 µg/Day + Sham
Started | 10 | 7
Completed | 5 | 6
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 1 | 1
Not completed — Study Terminated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients received either the 0.2µ/day or 0.5µ /day dose as well as a sham injection in the fellow eye. The total number of subjects enrolled/analyzed was 17.
Groups:
- A, 2, I 0.2 µg/Day + Sham: 0.2 µg/Day
  Fluocinolone Acetonide: 0.2 µg/Day + Sham treatment in fellow eye
- A, 2, II 0.5 µg/Day + Sham: 0.5 µg/Day
  Fluocinolone Acetonide: 0.5 µg/Day + Sham treatment in fellow eye
- Total: Total of all reporting groups
Arm/Group | A, 2, I 0.2 µg/Day + Sham | A, 2, II 0.5 µg/Day + Sham | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.95 (8.976) | 82.55 (6.056) | 81.02 (7.799)
Age, Customized [Number; unit: participants]
  <35 years | 0 | 0 | 0
  35-44 years | 0 | 0 | 0
  45-54 years | 0 | 0 | 0
  55-64 years | 1 | 0 | 1
  65-74 years | 1 | 1 | 2
  75-84 years | 5 | 2 | 7
  ≥85 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Size of Geographic Atrophy
Time Frame: 24 months
Population: Patients received either a 0.2µg/Day or 0.5 µg/Day treatment in the study eye and a sham treatment in the fellow eye.
Measure: Mean (Standard Deviation); unit: mm3/year
Groups:
- A, 2, I 0.2 µg/Day: 0.2 µg/Day
  Fluocinolone Acetonide: 0.2 µg/Day
- A, 2, II 0.5 µg/Day: 0.5 µg/Day
  Fluocinolone Acetonide: 0.5 µg/Day
Arm/Group | A, 2, I Sham | A, 2, I 0.2 µg/Day | A, 2, II Sham | A, 2, II 0.5 µg/Day
Number analyzed (Participants) | 8 | 8 | 6 | 6
mm3/year | 2.513 (1.5318) | 2.758 (1.7830) | 2.599 (2.4005) | 2.562 (1.9685)

ADVERSE EVENTS:
Description: Each patient received a sham injection in one eye and active treatment in the other eye.
Groups:
- Sham Injection: Sham Injection
  Sham Injection: Sham injection
  Ocular AEs
- 0.2 ug/Day: 0.2 µg/Day
  Fluocinolone Acetonide: 0.2 µg/Day
  Ocular AEs
- 0.5 ug/Day: 0.5 µg/Day
  Fluocinolone Acetonide: 0.5 µg/Day
  Ocular AEs
- 0.2 ug/Day + Sham Injection: Fluocinolone Acetonide: 0.2 µg/Day + Sham Injection
  Systemic AEs
- 0.5 ug/Day + Sham Injection: Fluocinolone Acetonide: 0.5 µg/Day + Sham Injection
  Systemic AEs
Arm/Group | Sham Injection | 0.2 ug/Day | 0.5 ug/Day | 0.2 ug/Day + Sham Injection | 0.5 ug/Day + Sham Injection
Serious Adverse Events (participants affected / at risk) | 3/17 | 3/10 | 2/7 | 3/10 | 5/7
Other Adverse Events (participants affected / at risk) | 10/17 | 8/10 | 7/7 | 5/10 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sham Injection (N=17) | 0.2 ug/Day (N=10) | 0.5 ug/Day (N=7) | 0.2 ug/Day + Sham Injection (N=10) | 0.5 ug/Day + Sham Injection (N=7)
Anaemia (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (2)
Renal mass (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 3 (3) | 3 (3) | 2 (2) | 0/0 (0) | 0/0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sham Injection (N=17) | 0.2 ug/Day (N=10) | 0.5 ug/Day (N=7) | 0.2 ug/Day + Sham Injection (N=10) | 0.5 ug/Day + Sham Injection (N=7)
Cardiac failure congestive (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Cataract (Eye disorders) | 3 (3) | 3 (4) | 2 (3) | 0/0 (0) | 0/0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Myodesopsia (Eye disorders) | 0 (0) | 2 (2) | 1 (2) | 0/0 (0) | 0/0 (0)
Photophobia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0)
Punctate keratitis (Eye disorders) | 5 (7) | 3 (3) | 3 (5) | 0/0 (0) | 0/0 (0)
Retinal pigment epithelial tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0)
Visual impairment (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Pneumonia (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 0/0 (0) | 0/0 (0)
Dehydration (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cutis laxa (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Phlebitis (Vascular disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days